CLINICAL TRIAL: NCT03812159
Title: Clinical Feasibility Study of Preoperative Surgical Planning for Craniosynostosis Procedures
Brief Title: Clinical Feasibility Study of Preoperative Surgical Planning
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study members relocated after Covid and recruitment stopped
Sponsor: Gary F. Rogers, MD (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor-Investigator, Gary F. Rogers, MD, Principal Investigator, Children's National Research Institute
Organization: Children's National Research Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00011015; R42HD081712 (NIH)
Record Dates: First submitted 2018-12-20; First posted 2019-01-23 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Craniosynostoses
Keywords: Shape analysis; Computer-assisted surgical plan; Surgical planning; Computational anatomy
MeSH Terms: conditions — Craniosynostoses

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Presurgical planning (Experimental): Undergo crania-vault reconstruction following the presurgical planning (iCSPlan)
  Interventions: Device: iCSPlan

INTERVENTIONS:
Device: iCSPlan — The Investigator will acquire a routine pre-operative CT-scan to help assess the synostosis severity. A week before the surgery a routine preoperative visit will be done. If the potential subject agrees to participate in the study, a presurgical plan will be built, and based on the CT scan, it will (1) quantify shape differences between pathological and healthy cranial shapes; (2) compensates for brain and cranial growth during the months between diagnosis, treatment and recovery; and (3) guides bone-cuts and bone-placement for the simplest and optimal surgical procedure.
  Finally this plan will be recorded in a software, iCSPlan, which will be reviewed by the surgeon. If it is accepted, it will be available during the surgery as a rely-on tool which may or may not be followed.

SUMMARY:
Most children diagnosed with craniosynostosis undergo a relatively extensive cranial vault remodeling procedure. The decision of performing surgical cranial shape correction for patients with craniosynostosis typically rests on a subjective visual assessment of the severity of the cranial malformation and the main goal of this procedure is to reduce the risk of elevated intracranial pressure and to provide a more normal cranial shape and volume. Personalized surgical planning systems to optimize intervention and leverage surgical expertise in the reconstruction of the cranial vault do not exist. Thus, the expertise of the surgeon is paramount for the success of the surgical correction of craniosynostosis. The goal of our project is to evaluate the feasibility and utility of a surgical plan derived from software developed at Children's National, iCSPlan.

DETAILED DESCRIPTION:
Presurgical planning will be performed in patients that require an open crania-vault reconstruction for craniosynostosis. The participants will come from the outpatient clinics of neurosurgery and plastic surgery. The treating physician/study team member will explain and give a copy of Institutional review board (IRB) approved study information letter to the participant's legally authorized representative (LAR).

The investigators will acquire a pre-operative CT-scan, per standard of care, to help assess the synostosis severity, within 4 weeks before the procedure. A week before the surgery, a routine preoperative visit will be done where the participant and/or LAR, if agree to participate in the study, will sign the informed consent document(s).

A presurgical plan will be built and will be recorded in a software, iCSPlan. Although this plan will not be integrated in the OR workflow, if needed, it would be visualized on a desktop monitor, which will be available to the surgical team. This tool will not influence any clinical decision making in the study. Instead, it will work as a rely-on tool in the preparation of the surgery, which may or may not be followed by the surgeon.

Demographic information (sex, age), as well as intraoperative information (Anesthesia length, anesthesia medications, length of surgery, blood loss, # of blood units transfused, complications), will be recorded for analysis. These variables are generally recorded during surgery and add no additional operative time.

Following the surgery, the specialists will evaluate the feasibility of the use of the presurgical plan by completing a questionnaire to report their options on (1): Quality of the surgical outcome; (2) the quality of the surgical strategy, and (3) the utility of the surgical planning in the treatment. The questions will be answered on a 5-point Likert scale, ranging from "not useful/strongly dislike" to "very useful/strongly like".

All study team pre-screening materials that contain participants information will be maintained on password protected computers. Only authorized study team members will have access to the pre-screening materials. Any pre-screening protected health information (PHI) that is collected will be destroyed once study enrollment is completed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients under 18 years of age.
2. Diagnosis of craniosynostosis.
3. Scheduled for open crania vault reconstruction.
4. Patients seen in Children's National Medical Center.

Exclusion Criteria:

1. Lack of interest in participating and refusal to consent.
2. Plan for endoscopic craniectomy of synostosis.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-03-20 (Estimated); Study Completion 2024-04-20 (Estimated)

PRIMARY OUTCOMES:
To evaluate the feasibility of a surgical planning software (iCSPlan) for open cranial vault reconstructions assessed by how often will the surgeon use or discard the surgical plan | a week before surgery
  Preoperative planning for cranial vault reconstruction will be built in patients under 18 years old with craniosynostosis. We will document the number of times the surgical plan is followed by the surgeon.

SECONDARY OUTCOMES:
To evaluate the utility of the surgical planning software (iCSPlan) assessed by a 5-point Likert scale questionnaire. | A week before surgery
  Surgeons will review the iCSPlan. To evaluate the utility of the plan, they will complete a questionnaire ranging from 1-5:
  1. Not at all useful;
  2. Slightly useful;
  3. Moderately useful;
  4. Very useful;
  5. Extremely useful.
To evaluate the quality of the surgical strategy and the surgical outcome built by the surgical planning software (iCSPlan) surgeons will complete a 5-point Likert scale questionnaire. | a week before surgery
  After reviewing the iCSPlan, surgeons will evaluate the quality of the surgical strategy and outcome by completing a questionnaire ranging from 1-5.
  1: Very poor 2. Poor 3. Fair 4. Good 5. Excellent
To evaluate the impact of the surgical planning software (iCSplan) assessed by the difference in the length of surgery if the plan is used. | The day of surgery (One day)
  Intra-operative variables such as time of surgery is a quantitative measure that would represent the effect of the use of the iCSPlan. We will compare this value in patients for whom the surgical plan was used and was not used.
To evaluate the intra-operative impact of using a surgical planning software (iCSPlan) assessed by the amount of blood loss, and thus, the amount of transfusion needed. | The day of surgery (One day)
  One of the major concern during an open cranial vault reconstruction is the amount of blood loss. Measuring this variable and the number of blood units transfused will let us evaluate the impact of the iCSPlan.
To evaluate the postoperative impact of undergoing a cranial vault reconstruction following the surgical planning software (iCSPlan) measured by the complications encountered 30-days after the surgery. | 30 days after surgery.
  Complications such as infection, bleeding, reintervention, brain injury, cranial bone loss, among others, will be recorded in a period of 30 days after the surgery. We will compare the number of complications encountered in patients for whom the surgical plan was used and was not used.
To evaluate the postoperative impact of undergoing a cranial vault reconstruction following the surgical planning software (iCSPlan) measured by the length of stay. | One month.
  We will compare the length of stay in patients for whom the surgical plan was used and was not used.

CONTACTS AND LOCATIONS:
Overall Officials: Gary Rogers, MD, Principal Investigator — Children's National Research Institute
Locations (1):
- Childrens National Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Porras AR, Paniagua B, Ensel S, Keating R, Rogers GF, Enquobahrie A, Linguraru MG. Locally Affine Diffeomorphic Surface Registration and Its Application to Surgical Planning of Fronto-Orbital Advancement. IEEE Trans Med Imaging. 2018 Jul;37(7):1690-1700. doi: 10.1109/TMI.2018.2816402. PMID 29969419
- [Background] Porras AR, Zukic D, Equobahrie A, Rogers GF, Linguraru MG. Personalized Optimal Planning for the Surgical Correction of Metopic Craniosynostosis. Clin Image Based Proced. 2016;2016:60-67. doi: 10.1007/978-3-319-46472-5_8. Epub 2016 Sep 21. PMID 28149960
- [Background] Porras AR, Paniagua B, Enquobahrie A, Ensel S, Shah H, Keating R, Rogers GF, Linguraru MG. Locally affine diffeomorphic surface registration for planning of metopic craniosynostosis surgery. Med Image Comput Comput Assist Interv. 2017 Sep;10434:479-487. doi: 10.1007/978-3-319-66185-8_54. Epub 2017 Sep 4. PMID 29527598